CLINICAL TRIAL: NCT03089762
Title: Intra-articular Injection in the Knee of Adipose Derived Stromal Cells and Platelet Rich Plasma for Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioheart, Inc. (Industry)
Collaborators: Anupam Hospital (Other); RegennMed Research and Therapeutics Delhi (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAH/02/12
Record Dates: First submitted 2017-03-15; First posted 2017-03-24 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SVF and PRP (Experimental)
  Interventions: Biological: Intra-articular injection of SVF plus PRP

INTERVENTIONS:
Biological: Intra-articular injection of SVF plus PRP — administering SVF and PRP intra-articularly into patients with osteoarthritis grade 1 and 2

SUMMARY:
Stromal vascular fraction (SVF) can easily be obtained from a mini-lipoaspirate procedure of fat tissue and platelet rich plasma (PRP) can be obtained from peripheral blood. Evaluated the safety and preliminary efficacy of administering SVF and PRP intra-articularly into patients with osteoarthritis grade 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* patients age 50 or older who present with symptomatic primary osteoarthritis of the knee
* daily pain for the previous 3 months
* analgesics usage at least once a week
* less than 30 minutes of morning stiffness
* WOMAC score of ≤ 75 in the target knee
* Brandt Radiographic Grading Scale of Osteoarthritis grade 1 and 2

Exclusion Criteria:

* evidence of secondary knee osteoarthritis
* severe osteoarthritis (Joint space width - JSW < 2 mm)
* prior intra articular injections within the previous one year prior to inclusion
* patients with clinically significant systemic disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02-12 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities Arthritis Index) | 1 year

SECONDARY OUTCOMES:
Six minute walk distance | 1 year

REFERENCES:
- [Derived] Bansal H, Comella K, Leon J, Verma P, Agrawal D, Koka P, Ichim T. Intra-articular injection in the knee of adipose derived stromal cells (stromal vascular fraction) and platelet rich plasma for osteoarthritis. J Transl Med. 2017 Jun 19;15(1):141. doi: 10.1186/s12967-017-1242-4. PMID 28629466 (Retraction: PMID 33902642 J Transl Med. 2021 Apr 26;19(1):168)